CLINICAL TRIAL: NCT01663428
Title: Sup-ER Splinting: Does Early Passive Positioning in Supination and External Rotation in Children With Birth Related Brachial Plexus Injury Have Benefit?
Brief Title: Sup-ER Splint for Children With Birth Related Brachial Plexus Injury
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: It was decided to change the study from a cohort to a randomized controlled trial.
Sponsor: University of British Columbia (Other)
Collaborators: Children's & Women's Health Centre of British Columbia (Other)
Responsible Party: Principal Investigator, Cynthia Verchere, Principle Investigator, University of British Columbia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H12-00776
Record Dates: First submitted 2012-08-09; First posted 2012-08-13 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Birth Related Brachial Plexus Injury; Obstetrical Brachial Plexus Palsy
Keywords: birth related brachial plexus injury; brachial plexus; splint
MeSH Terms: conditions — Neonatal Brachial Plexus Palsy | interventions — Splints

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sup-ER Splint (Experimental): Experimental group that will receive Sup-ER splint.
  Interventions: Other: Sup-ER Splint
- Control (Currently accepted treatment) (Active Comparator): Control group that will receive the currently accepted treatment.
  Interventions: Other: Currently accepted treatment

INTERVENTIONS:
Other: Sup-ER Splint
  Other Names: Splint
  Arms: Sup-ER Splint
Other: Currently accepted treatment
  Arms: Control (Currently accepted treatment)

SUMMARY:
This study evaluates the ability of a newly designed splint called "Sup-ER Splint" to improve the arm function and anatomy of children with birth related brachial plexus injuries.

DETAILED DESCRIPTION:
The brachial plexus is a group of 5 nerves from the spinal cord that provide the movement and sensation of an upper extremity. In some difficult deliveries, traction on the shoulder may lead to damage to the brachial plexus and will result in an arm that is paralyzed. This is called 'birth related brachial plexus injury' (BRBPI). This may occur in up to 1/1000 births and the nerves may be injured minimally to severely. About 2/3 of children with this injury will recover to quite functional levels simply by maintaining looseness of joints while their nerves slowly heal. Some children have nerve injuries severe enough that they require surgical reconstruction with nerve grafts and nerve transfers to achieve even adequate function. One almost universally common outcome, even in children with otherwise "good" recovery, is that the motions of external rotation of the shoulder and supination of the forearm are weaker, later to recover, and often incomplete. Even beyond these direct functional weaknesses, because the arm is positioned poorly, joint contractures and imbalance of these motions can interfere with other upper extremity movements like elbow flexion, even when elbow flexion itself is well recovered. More importantly, lack of full motion leads to long term changes in the structure, growth, and posture of the shoulder requiring further musculoskeletal surgery, or a child with permanent deformity or disability. Surgery cannot completely correct this deformity. Any gains in active and passive range of motion during the first year of life may improve these long-term shoulder outcomes. The investigators have instituted a program of early passive repositioning mostly using a custom Sup-ER (Supination and External Rotation) splint during early growth and development to improve arm position and range of motion where ER and Sup are weak. In compliant patients in a pilot study, the speed and strength of recovery of ER and Supination are improved compared to historical controls. It is a novel splint and protocol designed by the investigators and has significantly changed the care received by patients in BC. This study will evaluate the use of Sup-ER splint in multiple centres over a five year period by assessing the arm function at common time points in recovery.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of brachial plexus injury at birth.
* Significant deficit in external rotation and/or supination of the affected limb based on clinical assessment using the Toronto Active Movement Scale at 6 weeks of age: External Rotation ≤ 2 and/or Supination ≤ 2
* Tightness in Passive Range of Motion of external rotation: any angle of less than 180°.
* Age 6-8 weeks for complete protocol fulfillment.

Exclusion Criteria:

* Neuromuscular disorder.
* Unwillingness or inability to comply with the requirements of this protocol.

Ages: 6 Weeks to 8 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2012-07; Primary Completion 2015-08 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Toronto Active Movement Scale | 1 year of age

SECONDARY OUTCOMES:
Alpha angle (glenoid version) and posterior displacement of humeral head (PDHH) | 6 months of age
  The Alpha angle (glenoid version) and posterior displacement of humeral head (PDHH) will be measured at baseline and 6 months of age by ultrasound.

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Verchere, MD FRCSC, Principal Investigator — University of British Columbia